CLINICAL TRIAL: NCT04915443
Title: Periotome Versus Peizotome as an Aid of Atraumatic Extraction.
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Mohammed Alraqibah, Principal Investigator, Qassim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA/m-2019-3013
Record Dates: First submitted 2021-05-26; First posted 2021-06-07 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Dental Extraction; Dental Implant
Keywords: Extraction; Implant; Periotome; Piezotome; Atraumatic

STUDY DESIGN:
Intervention Model Description: All patients attending Qassim University dental clinics with teeth indicated for simple extraction will be assigned randomly to one of the two study groups either (Periotome Group) or (Piezotome Group) after insuring that they fit the inclusion criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Periotome Group (Experimental): An Atraumatic simple extraction procedure is done to teeth or roots with sound form indicated for simple extraction using H.ZEPF 26.182.13 & 26.182.11 periotome instrument.
  Interventions: Device: Periotome
- Piezotome Group (Experimental): An Atraumatic simple extraction procedure is done to teeth or roots with sound form indicated for simple extraction using SOLO LED PIEZOTOME Kit with ESSENTIAL tips from SATELEC ACTEON.
  Interventions: Device: Piezotome

INTERVENTIONS:
Device: Periotome — Dental instrument used to perform atraumatic dental extraction.
  After the initial de attachment, the periotome was inserted between the root and the bone parallel to the long axis of the root and pushed apically to the maximum depth that the tissue allowes severing the PDL and leaving it for 10-15 seconds allowing the biomechanical creep to occur.
  This proses is repeated at different points of entries at all the different surfaces of the tooth.
  Arms: Periotome Group
Device: Piezotome — Dental device used for many purposes one of which is performing atraumatic dental extraction.
  An LC2 tip was used for all the procedures and it was inserted between the tooth root and the bone parallel to the long axis of the root and moved in a sweeping motion 3-4mm toward the apex severing the PDL.
  Arms: Piezotome Group

SUMMARY:
This study aims to compare between periotome and piezotome in terms of efficiency and durability in procedures of simple extractions as an alternative atraumatic extraction technique.

DETAILED DESCRIPTION:
Teeth extraction is one of the commonly preformed procedures in the dental clinics, and one of the most important precautions followed during the different techniques of teeth extraction is tissue preservation and the avoidance of tissue trauma. So, for the preservation of bone and tissues integrity and elimination of post operative pain and discomfort, atraumatic extraction techniques are presented.

A claim has risen that due to its thin tips which is inserted vertically to the PDL avoiding the leveraging forces caused by conventional elevators, Periotome will aid in the reduction of soft tissue injury and the preservation of bone integrity. While Piezotome which is a newer and innovative device using ultrasonic vibrations mainly for the purpose of osteotomy is considered very efficient due to its selective cutting and being inert against soft tissues, including nerves and blood vessels. leading to lesser cell necrosis and faster bone regeneration providing a minimally invasive atraumatic extraction technique.

And with the rapid development of implantology and painless dentistry, the demands on more efficient, minimally invasive and more durable atraumatic extraction techniques has increased.

This study aims to compare between periotome and piezotome in terms of efficiency and durability in procedures of simple extractions as an alternative atraumatic extraction technique.

ELIGIBILITY:
Inclusion Criteria:

* Grade I or II patients according to ASA
* Teeth indicated for simple extraction
* Teeth indicated for extraction and immediate implant placement
* Teeth of grade 0-I Mobility
* Remaining roots with sound form

Exclusion Criteria:

* Grade III-VI patients according to ASA
* Mobility Grade ≥ II
* Teeth indicated for surgical extraction

  * ASA: American Society of Anesthesiologists Physical Status Classification System 2020

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Operative Duration | From the beginning of extraction tell the delivery of the tooth out from the socket. From the beginning of intervention up to 60 minutes
  To compare the operative duration of simple extraction between "Periotome" and "Piezotome" in (minutes).
Gingival Laceration | At the end of the extraction procedure up to 60 minutes
  To identify the presence or absence of gingival laceration in the extraction area Immediately after the completion of the extraction procedures (yes/no).
Operative Pain | From the beginning of extraction tell the delivery of the tooth out from the socket. From the beginning of intervention up to 60 minutes
  To evaluate operative pain felt by the patient during the two procedures using (visual analogue scale). The patient is asked after the procedure to give a pain score (using visual analogue scale) to evaluate his/her pain during the procedure.
  0= no pain (best outcome) 10= unberable pain (worst outcome)
Post-Operative Pain | 8 hours following the Procedure tell the 7th day.
  To evaluate post-operative pain felt by the patient after the two procedures using (visual analogue scale). The patient is asked after the procedure to give a pain score (using visual analogue scale) to evaluate his/her pain following the procedure in the following order: (1st day, 2nd day, 3rd day and 7th day) from the completion of the procedure.
  0= no pain (best outcome) 10= unberable pain (worst outcome)
Analgesics Intake | 8 hours following the intervention tell the 7th day.
  To calculate the dosage (in mg) of analgesics intake by the patient after the two procedures. The patient is asked to record his/her analgesics intake daily by dose and in the first 7 days following the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: DAYASHANKARA JK RAO, MDS,MFDSRCS, Study Director — College of Dentistry Qassim University, Kingdom of Saudi Arabia
Locations (1):
- Qassim Unversity Dental Clinics, Buraidah, Saudi Arabia

REFERENCES:
- [Background] Srivastava P, Shetty P, Shetty S. Comparison of Surgical Outcome after Impacted Third Molar Surgery Using Piezotome and a Conventional Rotary Handpiece. Contemp Clin Dent. 2018 Sep;9(Suppl 2):S318-S324. doi: 10.4103/ccd.ccd_354_18. PMID 30294165
- [Background] Malden N. Surgical forceps techniques. Dent Update. 2001 Jan-Feb;28(1):41-4. doi: 10.12968/denu.2001.28.1.41. PMID 11819949
- [Background] Sharma SD, Vidya B, Alexander M, Deshmukh S. Periotome as an Aid to Atraumatic Extraction: A Comparative Double Blind Randomized Controlled Trial. J Maxillofac Oral Surg. 2015 Sep;14(3):611-5. doi: 10.1007/s12663-014-0723-8. Epub 2014 Nov 8. PMID 26225052
- [Background] Bhati B, Kukreja P, Kumar S, Rathi VC, Singh K, Bansal S. Piezosurgery versus Rotatory Osteotomy in Mandibular Impacted Third Molar Extraction. Ann Maxillofac Surg. 2017 Jan-Jun;7(1):5-10. doi: 10.4103/ams.ams_38_16. PMID 28713729
- [Background] Chang HH, Lee MS, Hsu YC, Tsai SJ, Lin CP. Comparison of clinical parameters and environmental noise levels between regular surgery and piezosurgery for extraction of impacted third molars. J Formos Med Assoc. 2015 Oct;114(10):929-35. doi: 10.1016/j.jfma.2014.02.003. Epub 2014 Mar 21. PMID 24661578

DOCUMENTS (1):
  • Informed Consent Form (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT04915443/ICF_000.pdf